CLINICAL TRIAL: NCT01973920
Title: A Single Center, Multiple-dose, Non-randomized, Dose Adjustment, Open-Label Study to Evaluate the Efficacy, Pharmacodynamics, Safety, and Tolerability of Oshadi Icp in Patients With Type 1 Diabetes Mellitus -A Phase II Clinical Study
Brief Title: Efficacy Safety and Tolerability of Multiple Doses of Oshadi Icp (Oshadi Oral Insulin) in Patients With Type 1 Diabetes Mellitus - Phase II Clinical Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oshadi Drug Administration (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OS-ICP-P2 -01
Record Dates: First submitted 2013-10-27; First posted 2013-11-01 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2016-03

CONDITIONS: Diabetes Mellitus; Insulin-Dependent; Type 1
Keywords: Diabetes Mellitus; Oral Insulin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

ARMS (1):
- Oshadi Icp (Experimental): Oshadi Icp oral insulin,
  Interventions: Drug: Oshadi Icp

INTERVENTIONS:
Drug: Oshadi Icp
  Other Names: Oral insulin

SUMMARY:
Diabetes mellitus (DM) is a chronic disease of carbohydrate, fat, and protein metabolism caused by an absolute or relative deficiency of insulin, an anabolic hormone. The current methods of insulin therapy for diabetic patients are multiple daily injection therapy and continuous subcutaneous insulin infusion with an external pump. This rout of administration may lead to hyperinsulinemia as insulin is administered in a non physiological way, targeting mainly extra hepatic tissues (muscle, fat). A method of providing insulin without the need for injections has been a goal in drug delivery.

Oshadi Drug Administration Ltd. has developed oral carrier for proteins based on biochemistry and quantum theory of biochemical reactions. The carrier enables the absorption of proteins from the gastrointestinal tract in their full structure. Oshadi has also developed the Oshadi Icp - insulin, proinsulin and C-peptide in Oshadi carrier, administrated orally. This study was design in order to evaluate the safety and feasibility of multiple administrations of Oshadi Icp for home use. The study will be a multiple-dose, open-label non-randomized study in patients with Type 1 diabetes, with periodic dose adjustments. The study will include 4 weeks of multiple-dose administration of Oshadi oral insulin (Oshadi Icp) at home and in study center for the determination of the efficacy, safety and pharmacodynamic effects of Oshadi Icp.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (according to ADA criteria) for more than 3 year.
* Male/female 21 years old and older.
* BMI≥18.5 and ≤25
* Female of childbearing age must commit to avoid pregnancy and use contraception during the study.
* Patients must understand and be willing to give written informed consent prior to any study procedures or evaluations and be willing to adhere to all study schedules and requirements.

Exclusion Criteria:

* Any history of significant cardiac, renal, neurologic, metabolic, pulmonary, gastrointestinal, hematologic abnormality, chronic hepatic disease or any other disease which in the judgment of the investigator would interfere with the study or confound the results.
* Symptomatic DKA (diabetic ketoacidosis)in the last 6 months
* Patients with positive HIV or HCV (hepatitis C virus)serology or positive HBsAg at screening.
* History or evidence of any active liver disease.
* History of epilepsy.
* One or more episodes of sever hypoglycemia during the last 12 months
* History of hypoglycemic unawareness.
* C-peptide >3 mg/ml (fasting)
* Total average daily insulin dosage ≥1 IU/kg of body weight.
* Polycystic ovary syndrome
* Acanthosis nigricans
* 6.5% > HbA1c or HbA1c >10%
* eGFR<60 (epidermal growth factor receptor).
* Female patients who are breastfeeding or have a positive pregnancy test at screening or at any time during the study and not willing to practice birth control during study period.
* Inability to give written informed consent
* History of alcohol or drug abuse within 6 months of screening.
* Patients who have a positive urine drug screen for substances of abuse (benzodiazepine, THC (tetrahydrocannabinol), opiates, amphetamines, cocaine) at the screening.
* Mental disorders.
* Significant swallowing disorders
* Digestive disorders
* Small bowel surgery
* Any intercurrent disease during the last week prior to screening which in the judgment of the investigator might affect blood glucose level.
* Any infectious disease developed during the 4 weeks prior to the study.
* Malabsorption disorders.
* Any significant abnormality by principal investigator in the baseline laboratory evaluation: liver and kidney functions, electrolytes, albumin, lipase, TSH (thyroid-stimulating hormone), hemoglobin, white blood cell count and differential, platelets.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events occurence | last follow-up visit (day 60)

SECONDARY OUTCOMES:
To assess the pharmacodynamic effect of multiple doses of Oshadi Icp as measured by the area under the glucose concentration-time curve | Last administration day (day 37)

OTHER OUTCOMES:
Evaluating the total daily injected insulin dose during administration of Oshadi Icp vs routine use | Last administration day (day 37)

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Rachmiel, Dr., Principal Investigator — Assaf-Harofeh Medical Center, Israel
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel